CLINICAL TRIAL: NCT02530853
Title: Acupuncture as Applied Technology to Nursing Care Adult Hypertensive: An Experimental Study.
Brief Title: Acupuncture as a Complementary Treatment for Hypertension (ACT-HAS)
Acronym: ACT-HAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Collaborators: Ministry of Health, Brazil (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, NEIDE APARECIDA TITONELLI ALVIM, PhD, Nurse, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 32909414.4.1001.5238; 772.508 (Other: Nº do Parecer do CEP)
Record Dates: First submitted 2015-08-19; First posted 2015-08-21 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Hypertensive Disease
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): Laser acupuncture
  Interventions: Other: Laser acupuncture
- Group B (Sham Comparator): Simulation Laser acupuncture
  Interventions: Other: Laser acupuncture

INTERVENTIONS:
Other: Laser acupuncture — Laser acupuncture

SUMMARY:
This is a randomized clinical trial with blinded, multi-center, involving the Federal University of in Rio de Janeiro(UFRJ), through the School of Nursing Anna Nery, as a proponent and research coordinator; and as a collaborative educational institutions, the Federal University of in Espirito Santo, represented by the Department of Nursing; and the Higher School of Sciences of the Santa Casa de Misericordia of Vitoria, developed by building doctorate thesis as a final product of the research.

DETAILED DESCRIPTION:
The objective of investigation is the effectiveness of acupuncture as a complementary health care to patients with primary hypertension drug therapy.

Methodological approach - Randomized Clinical Trial triple blind.

Population / sample - Patients with Primary Hypertension in drug treatment for over a year and no effective control of blood pressure levels, that is, regular saving measures above was over 140x90 mmHg.

How centers Participants Research, the study covers health units of the Municipal Health of Maricá in Rio de Janeiro, the Municipal of Victoria Health in Espirito Santo, beyond the scope of Integrated Project Research-Service (PIPA), linked to School Nursing Anna Nery /UFRJ.

Primary Objective - To evaluate the effectiveness of acupuncture as a complementary health practice associated with drug treatment used in adults with primary hypertension, based on nursing diagnoses.

Secondary objectives:

* Estimate blood pressure levels after exposure to acupuncture applied in adults with primary hypertension.
* Draw the profile of the most frequent nursing diagnoses in adults with primary hypertension.
* Analyze the effectiveness of acupuncture as a complementary health therapy associated with drug treatment used on these clients, based on nursing diagnoses.

ELIGIBILITY:
Inclusion Criteria:

* Be suffering from essential hypertension;
* Be properly prescribed medication and have difficulty controlling blood pressure keeping regular measurement above was over 140x90 mmHg.

Exclusion Criteria:

* A woman in pregnancy;
* Be in possession of any type of cancer;
* being a smoker;
* be alcoholic;
* Be in drug treatment for other diseases including obesity;
* Not dieting for weight loss;
* practice regular physical activity.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-12 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Improvement of blood pressure levels. | six weeks

SECONDARY OUTCOMES:
Improvement of nursing diagnoses | six weeks

CONTACTS AND LOCATIONS:
Overall Officials: Neide Alvim, Study Director — UFRJ; Claudia Pereira, Study Chair — UFRJ
Locations (1):
- Raphael, Rio de Janeiro, Maricá, Brazil

REFERENCES:
- [Derived] Pereira RDM, Alvim NAT, Pereira CD, Gomes Junior SCDS. Laser acupuncture protocol for essential systemic arterial hypertension: randomized clinical trial. Rev Lat Am Enfermagem. 2018 Jul 16;26:e2936. doi: 10.1590/1518-8345.1887.2936. PMID 30020330